CLINICAL TRIAL: NCT07196826
Title: Effect of Passive Versus Active Aquatic Therapy Over Conventional Physiotherapy in Patients With Chronic Low Back Pain - A Randomized Crossover Trial
Brief Title: Effect of Passive Versus Active Aquatic Therapy Compared With Conventional Physiotherapy for Chronic Low Back Pain
Acronym: AQUA-LBP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-COHS-STD-122-APR-2024
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Aquatic Therapy (Experimental): Participants perform exercises in water, actively moving their back, core, and legs. The buoyancy of water reduces stress on the spine and joints, making movements easier and safer. This therapy focuses on improving strength, flexibility, core stability, balance, and overall function. Each session is guided by a licensed physiotherapist who ensures proper technique and monitors participants for safety. This approach aims to reduce chronic low back pain, improve mobility, and enhance daily activity performance and quality of life.
  Interventions: Procedure: Active Aquatic Therapy
- Passive Aquatic Therapy (Experimental): Participants receive assisted movements in water guided by a trained physiotherapist. The therapist moves the participant's back, core, and legs gently, allowing for improved spinal mobility, reduced stiffness, and relaxation without stressing the lower back. Water resistance and support help increase flexibility and reduce pain. Each session is supervised to ensure safety, correct technique, and comfort. This method aims to relieve chronic low back pain, improve function, and enhance participants' ability to perform daily activities safely and comfortably.
  Interventions: Procedure: Passive Aquatic Therapy
- Conventional Physiotherapy (Active Comparator): Participants perform standard land-based exercises including stretching, strengthening, and core stabilization exercises under the supervision of a licensed physiotherapist. The therapy focuses on improving spinal mobility, core strength, posture, and functional ability, aiming to reduce pain and improve daily activities. Each session is tailored to the participant's abilities and monitored for safety and correct technique. This conventional physiotherapy serves as the standard comparator to evaluate the effectiveness of aquatic therapies in managing chronic low back pain and enhancing quality of life.
  Interventions: Procedure: Conventional Physiotherapy

INTERVENTIONS:
Procedure: Active Aquatic Therapy — Active Aquatic Therapy involves structured, therapist-guided exercises in a heated hydrotherapy pool (32-34°C). Water buoyancy and resistance reduce spinal load, facilitate movement, and enhance muscle activation. Sessions last 45-60 minutes, 3 times per week for 4 weeks, supervised by licensed physiotherapists. Each session includes warm-up (water marching, arm swings, trunk rotations), main exercises (lumbar spine function, core strengthening, balance, hip abduction, back extensions, aqua walking, arm/leg strengthening), and cool-down (floating, deep breathing, passive stretches). Intensity is monitored using the Borg RPE scale (60-80% max HR). This intervention uniquely uses active engagement in water to reduce pain and improve strength, flexibility, and function, distinguishing it from passive aquatic therapy and land-based physiotherapy.
  Arms: Active Aquatic Therapy
Procedure: Passive Aquatic Therapy — Passive Aquatic Therapy (Watsu) is a therapist-guided, passive aquatic technique performed in a warm hydrotherapy pool (35°C). The patient floats while the therapist gently moves their body in rhythmic, synchronized patterns, providing massage, stretching, joint mobilization, and acupressure. Sessions last 45-60 minutes, 3 times per week for 4 weeks, and include preparation/floating, cradling with passive movements, passive stretching and mobilization, acupressure, and final relaxation. Neck and knee supports are used for comfort. This intervention uniquely emphasizes passive relaxation and gentle mobilization, making it suitable for patients with severe movement limitations, distinguishing it from active aquatic therapy and conventional land-based physiotherapy.
  Arms: Passive Aquatic Therapy
Procedure: Conventional Physiotherapy — Conventional Physiotherapy is a land-based intervention for chronic low back pain, delivered in an outpatient physiotherapy clinic. Sessions last 45 minutes, 3 times per week for 4 weeks, and include hot pack application (10-12 min) to reduce stiffness, electrotherapy (TENS/Interferential, 15 min) for pain modulation, and supervised therapeutic exercises (15-20 min) focusing on lumbar mobility, core stability, and spinal strengthening. Exercises include William's flexion, prone press-ups, cat-cow mobilization, hamstring stretches, pelvic tilts, and abdominal bracing. This intervention emphasizes pain reduction, postural control, and strengthening deep abdominal and paraspinal muscles, distinguishing it from passive and active aquatic therapies, and serves as the standard comparator in this crossover study.
  Arms: Conventional Physiotherapy

SUMMARY:
This study is designed to help people with chronic low back pain, which is pain in the lower back that persists for more than three months and can affect daily life, including sitting, standing, walking, lifting, and other routine activities. Chronic low back pain can also impact work, mood, and overall quality of life, making it important to find effective rehabilitation methods that reduce pain and improve function.

The study compares the effects of three different rehabilitation approaches:

1. Active aquatic therapy - participants perform exercises in water where they actively move their back, core, and legs. The water helps support the body and reduces stress on the spine, allowing safer and easier movement. This approach aims to improve strength, flexibility, core stability, and overall function.
2. Passive aquatic therapy - participants receive assisted movements in water guided by a trained physiotherapist. This gentle method helps increase spinal mobility, reduces stiffness, promotes relaxation, and can relieve pain without placing stress on the lower back.
3. Conventional physiotherapy - participants perform standard exercises on land, including stretching, strengthening, and core stabilization exercises. All sessions are supervised by licensed physiotherapists to ensure exercises are done safely and effectively.

Participants will be randomly assigned to one of the three groups. Each intervention lasts 4 weeks, with multiple sessions each week. All sessions are supervised to provide proper guidance, ensure safety, and adapt exercises to each participant's needs.

Before starting therapy, participants' pain levels, core strength, flexibility, spinal mobility, and ability to perform daily activities will be measured using simple and understandable assessments. These measures will be repeated at the end of the 4-week intervention to evaluate improvements and compare the effectiveness of each rehabilitation approach.

The study is safe and non-invasive. No surgery, injections, or medications are involved. Participants' personal information is kept confidential, and all collected data will be used solely for research purposes.

By participating in this study, patients may benefit from structured, supervised rehabilitation that could help reduce pain, improve mobility and strength, enhance balance and core stability, and increase confidence in performing daily activities. Patients' feedback during sessions will also help researchers understand their experiences and preferences, which can improve future treatment recommendations.

The results of this study will help patients, families, physiotherapists, and healthcare providers understand which type of rehabilitation is most effective for chronic low back pain. This information can guide treatment decisions, improve individualized care plans, and support patients in returning to normal activities with less discomfort and greater independence.

Overall, the study aims to provide clear, practical information about rehabilitation options for chronic low back pain, improve functional outcomes, and enhance quality of life. Participants' contributions will help generate evidence that may benefit others with similar conditions in the future, while also receiving safe and professional care throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 65 years.
* Diagnosed with nonspecific chronic low back pain (duration >3 months).
* Capable of attending sessions and providing written informed consent. -

Exclusion Criteria:

* Acute low back pain or red flags (fractures, malignancy, infection).
* Recent spinal surgery (<6 months).
* Neurological disorders affecting balance or gait.
* Cardiopulmonary conditions contraindicating immersion.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Measured at baseline (before any intervention) and after each 4-week intervention phase.
  Pain intensity will be assessed using the Visual Analog Scale (VAS, 0-10 cm), where participants indicate their current level of low back pain from "no pain" to "worst imaginable pain." The VAS is a validated and reliable tool with high internal consistency and test-retest reliability.
  Purpose: To measure change in pain intensity associated with chronic low back pain.

SECONDARY OUTCOMES:
Functional Disability Oswestry Disability Index (ODI) | Measured at baseline and after each 4-week intervention phase.
  The ODI assesses limitations in daily activities due to low back pain, including sitting, standing, walking, and lifting. The instrument demonstrates excellent internal consistency (Cronbach's α = 0.82-0.90) and high reliability (ICC = 0.90-0.96).
  Purpose: To measure change in functional disability related to low back pain.
Lumbar Range of Motion (ROM) | Measured at baseline and after each 4-week intervention phase.
  Lumbar ROM will be measured using a double inclinometer according to AMA guidelines. Flexion and extension measurements are used to assess spinal mobility and functional flexibility. This method demonstrates high reliability for lumbar movement assessment.
  Purpose: To measure change in lumbar flexibility and range of motion.

CONTACTS AND LOCATIONS:
Locations (1):
- Gulf medical University, Ajman, Al Jurf, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided